CLINICAL TRIAL: NCT06602934
Title: Long-term Alterations of Host-microbiome Interactions and Cardiovascular and Respiratory Diseases Progression After Pneumonia - the HOMI-LUNG Project - Hospital-Acquired-Pneumonia
Brief Title: Long-term Alterations of Host-microbiome Interactions and Cardiovascular and Respiratory Diseases Progression After Pneumonia
Acronym: HOMI-LUNG-HAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC24_0112
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Hospital Acquired Pneumonia (HAP); Cardiovascular and Respiratory Disease
Keywords: Hospital-acquired pneumonia; Cardiovascular and respiratory diseases; Respiratory microbiome
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Respiration Disorders; Respiratory Tract Diseases | interventions — Blood Specimen Collection; Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A : Patients with acute major cardiovascular event (Other): Comparator
  Interventions: Other: Blood samples; Other: Oropharyngeal swabs; Other: Calcium score (CT scan); Other: ECG; Other: Cardiopulmonary exercise test, spirometry, plethysmography, pulmonary absorption of carbon monoxide in a single inspiration, and 6-minute walk test
- Group B: Patients with severe chronic cardiovascular disease (Other): Comparator
  Interventions: Other: Blood samples; Other: Oropharyngeal swabs; Other: Calcium score (CT scan); Other: ECG; Other: Cardiopulmonary exercise test, spirometry, plethysmography, pulmonary absorption of carbon monoxide in a single inspiration, and 6-minute walk test
- Group C: Patients with a high risk of CVD, yet no known history of CVRD or HA (Other): Comparator
  Interventions: Other: Blood samples; Other: Oropharyngeal swabs; Other: Calcium score (CT scan); Other: ECG; Other: Cardiopulmonary exercise test, spirometry, plethysmography, pulmonary absorption of carbon monoxide in a single inspiration, and 6-minute walk test
- Group D: Patients cured of HAP (Experimental)
  Interventions: Other: Blood samples; Other: Oropharyngeal swabs; Other: Calcium score (CT scan); Other: ECG; Other: Cardiopulmonary exercise test, spirometry, plethysmography, pulmonary absorption of carbon monoxide in a single inspiration, and 6-minute walk test

INTERVENTIONS:
Other: Blood samples — Four blood samples will be taken outside standard care for groups A, B, C and D: at inclusion, M6, M18 and M30 (only at inclusion for group C).
Other: Oropharyngeal swabs — An oropharyngeal swab will be taken to analyze patients' upper airway microbiome at inclusion, M6, M18 and M30.
Other: Calcium score (CT scan) — A calcium score will be taken at 30 months, to assess individual cardiovascular risk.
Other: ECG — Performed at inclusion, M6, M18 and M30
Other: Cardiopulmonary exercise test, spirometry, plethysmography, pulmonary absorption of carbon monoxide in a single inspiration, and 6-minute walk test — Cardiopulmonary exercise test, spirometry, plethysmography, pulmonary absorption of carbon monoxide in a single inspiration, and 6-minute walk test: These tests will be performed consecutively for 2 hours at inclusion (6-minute walk test only), at M6 and at M30. These tests will be performed to assess respiratory and cardiac function.

SUMMARY:
The HOMI-LUNG - HAP study is part of the HOMI-LUNG project, funded by the Horizon Europe program. The "HOMI-LUNG" project is an international, interdisciplinary project that aims to better understand the causal links between respiratory tract infections (i.e. pneumonia) and the progression of cardiovascular disease. More specifically, the project aims to quantify the burden of cardiovascular disease after pneumonia and assess patients' acceptability of long-term health alterations, as well as to define pneumonia endotypes with distinct pathobiological mechanisms associated with exacerbation of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

Group A (patients with acute cardiac disease)

* Male or female
* Age ≥ 40years old
* Hospitalized for acute coronary syndrome for less than 7 days.
* Informed consent from the patient
* Person insured under a health insurance scheme

Group B (patients with chronic cardiovascular disease)

* Male or female,
* Age ≥ 40 years old
* Undergoing coronary artery by-pass surgery
* Hospitalized in intensive care unit for > 12 hours
* Informed consent from the patient
* Person insured under a health insurance scheme

Group C (patients at risk of CVRD without chronic cardiovascular disease)

* Male or female,
* Age ≥ 40 years old
* Familial high levels of cholesterol or triglycerides
* With no personal history of CVRD, with a recent negative cardiac exercise test (last test inferior to 12 months)
* Follow-up for lipid abnormalities at high risk of CVRD events
* Informed consent from the patient
* Person insured under a health insurance scheme

Group D (patients with HAP)

* Male or female
* Age ≥ 40years old
* With one or more risk factors for CVD among:

smoking, abnormal lipidic levels, high blood pressure, obesity, diabetes mellitus, chronic kidney disease

* Cured from mechanically ventilated HAP during the current hospitalization
* Informed consent from the patient or relatives
* Person insured under a health insurance scheme

Exclusion Criteria:

* o Groups A, B, C and D
* Age >80 years old
* Immunosuppression pre-existing to the index hospitalisation, defined as lymphopenia < 500 elements/mm3, haematologic cancer, aplasia, chemotherapy/radiotherapy for cancer within 3 months prior to the inclusion, or anti-graft rejection drug.
* Pregnant women, breastfeeding women.
* Adults under guardianship or trusteeship.
* Low probability of survival at day 28.

  o Groups A, B, C
* Community-acquired pneumonia or Hospital-acquired pneumonia within the last year.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2029-01-02 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 6 months
  Major adverse cardiovascular events (MACE) at 6 months
Poor cardiorespiratory fitness | 30 months
  Poor cardiorespiratory fitness at 30 months. Poor tolerance is a VO2max lower than normal values for age

SECONDARY OUTCOMES:
Health care costs of CVRD progression after HAP | 18 months
  Health care costs of CVRD progression after HAP over 18 months
Rate of events | Month 6 and Month 30
  Rate of events : nonfatal stroke, nonfatal myocardial infarction, hospital admission for heart failure, and cardiovascular death
Rate of thrombo-embolic events | Month 6 and Month 30
  Rates of thrombo-embolic events : pulmonary embolism, deep venous thrombosis
Rates of CVD | Month 6 and Month 30
  Rates of CVD
Rates of major respiratory events | Month 6 and Month 30
  Rates of major respiratory events are defined as COPD exacerbation, asthma exacerbation, hospitalization for respiratory failure, and respiratory-related mortality at 6 and 30 months
NYHA (New York Heart Association) classification | Month 6, Month 18 and Month 30
  NYHA (New York Heart Association) classification of dyspnea
mMRC (Modified Medical Research Council) Dyspnoea Scale | Month 6, Month 18 and Month 30
  mMRC (Modified Medical Research Council) Dyspnoea Scale (Grade O to 4 : grade O = I only get breathless with strenuous exercise ; grade 4 : I am too breathless to leave the house or I am breathless when dressing/undressing)
Rate of restrictive chronic respiratory distress | Month 6 and Month 30
  Rate of restrictive chronic respiratory distress defined as% of patients withCPT (Total Lung Capacity) lower than normal values
Rate of obstructive chronic respiratory distress progression | Month 6 and Month 30
  Rate of obstructive chronic respiratory distress progression
Percentage of patients with diffusion capacity for carbon monoxide (DLCO) lower than normal values for age and sex | Month 6 and Month 30
  Percentage of patients with diffusion capacity for carbon monoxide (DLCO) lower than normal values for age and sex
Percentage of patients with vital capacity, expiratory reserve volume, and inspiratory reserved volume lower than normal values for age and sex | Month 6 and Month 30
  Percentage of patients with vital capacity, expiratory reserve volume, and inspiratory reserved volume lower than normal values for age and sex
Rate of patients with secondary lower respiratory tract infection | Month 6 and Month 30
  Rate of patients with secondary lower respiratory tract infection defined as clinical signs of infection with new infiltrate on Chest-X-Ray
Rate of patients with non-respiratory infection | Month 6 and Month 30
  Rate of patients with non-respiratory infection
Rates of patients with the Montreal Cognitive Assessment (MoCA) score values lower than 27 | Month 6 and Month 30
  Rates of patients with the Montreal Cognitive Assessment (MoCA) score values lower than 27 at M6 and at M30
Glasgow Outcome Scale Extended values | Month 6 and Month 30
  Glasgow Outcome Scale Extended values to assess global disability and recovery after traumatic brain injury
Brief Pain Inventory score | Month 6, Month 18 and Month 30
  BPI score. This self-assessment questionnaire assesses the maind imensions of pain : intensity, functional disability, social and family repercussions and level of psychological distress (scale 0-10 : 0 = no pain , 10 = worst pain)
Rates of patients with chronic pain | Month 6, Month 18 and Month 30
  Rates of patients with chronic pain (yes/no) as defined as worse pain score value within the last 24 hours superior to 3
Rates of patients with severe symptoms of anxiety | Month 6, Month 18 and Month 30
  Rates of patients with severe symptoms of anxiety defined as HADS_A greater than or equal to 11
Mean Satisfaction With Life Scale (SWLS) score | Month 6, Month 18 and Month 30
  Experience of CVRD progression from the patients' perspectives assessed by mean SWLS score
Correlation between SWLS and EQ-5D-5L dimensions and utility scores | Month 6, Month 18 and Month 30
  Correlation between Satisfaction With Life Scale (SWLS) and 5-level EQ-5D dimensions and utility scores
SF(Short Form)-36 score | Month 6, Month 18 and Month 30
  Patients' responses to the SF-36 at months 6, 18 and 30 in order to estimate the change in Health-Related Quality of Life (HRQoL) over time
Fatigue Severity Scale | Month 6, Month 18 and Month 30
  Patients' responses to the Fatigue Severity Scale at month 6, 18 and 30 in order to estimate change in perceived fatigue over time
Mean QALYs (Quality-Adjusted Life-Years) | 30 months
  Mean QALYs (Quality-Adjusted Life-Years) at 30 months
EPICES (Evaluation of precariousness and health inequalities in health examination centers) score | Month 6, Month 18 and Month 30
  Rate of socio-economical precarity defined as EPICES (Evaluation of precariousness and health inequalities in health examination centers) score values > 30 at M6, 18 and M30
Modelisation of host-microbiome interactions | Month 0, Month 6, Month 18 and Month 30
  Modelisation of host-microbiome interactions
CVD progression | Month 6 and Month 30
  CVD progression at Month 6 and Month 30

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Angers University Hospital, Angers
  - Nantes University Hospital, Nantes
  - Rennes University Hospital, Rennes
  - Rouen University Hospital, Rouen
  - Toulouse University Hospital, Toulouse